CLINICAL TRIAL: NCT04154722
Title: Treatment of 21st Century Typhoid Fever in Children;Open Label Mono vs Combination Drug Therapy
Brief Title: Comparison of Two Drugs Regimen in Treatment of Complicated Typhoid Fever in Children
Acronym: [XDRTYPHOID]
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ziauddin University (Other)
Responsible Party: Principal Investigator, Dr. Fatima G Siddiqi, MD resident, Ziauddin University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0980419HRPED
Record Dates: First submitted 2019-11-04; First posted 2019-11-06 (Actual); Last update posted 2021-06-16 (Actual); Status verified 2021-06

CONDITIONS: Typhoid Fever
Keywords: XDR TYPHOID FEVER
MeSH Terms: conditions — Typhoid Fever | interventions — Meropenem

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- meropenum and azithromycin group (Experimental): inj meropenum 20mg/kg/dose I/v in 3 divided doses and syp azithromycin 20mg/kg/day in 2 divided doses.
  Interventions: Drug: Meropenem Injection; Drug: Azithromycin Powder
- meropenum group (Active Comparator): inj meropenum 20mg/kg/dose I/v in 3 divided doses
  Interventions: Drug: Meropenem Injection

INTERVENTIONS:
Drug: Meropenem Injection — inj meropenum for 10 days
  Other Names: meroneum; penro
Drug: Azithromycin Powder — syp azithromycin for10days
  Other Names: azomax; zetro
  Arms: meropenum and azithromycin group

SUMMARY:
This study evaluates whether XDR Typhoid fever in children can be effectively treated with monotherapy (meropenum alone), or a combination (meropenum and azithromycin).

DETAILED DESCRIPTION:
Complicated XDR Enteric fever is a very serious systemic disease, caused by an extremely resistant mutant strain of Salmonella Typhi ( the H58 S. Typhi superbug,) that as the name suggests is resistant to not only the first but also the second tier drugs conventionally used for treatment of the same. And as such, warrants immediate antibiotic therapy, but in view of the extended antimicrobial resistance the treatment options are limited to only two effective drugs viz Carbepenem and Azithromycin, as per culture sensitivity.

So far, in the absence of universal standardized treatment protocols for XDR complicated typhoid fever in children, random use of either one or both in combination is the current practice.

However, keeping antibiotic stewardship in mind, it is imperative to ascertain whether meropenum alone is effective or should be combined with azithromycin in the treatment of this serious disease.

Our study therefore compares the efficacy of monotherapy with meropenum or combination with azithromycin based on clinical and microbiologic remission, shortened hospital stay and less chances of relapse in order to then formulate a standardized protocol to treat complicated XDR typhoid in children thus preventing yet further antimicrobial resistance.

ELIGIBILITY:
Inclusion Criteria:

Patients with extended drug resistant typhoid fever defined as culture proven typhoid fever caused by Salmonella Typhi or Para typhi resistant to Ampicillin, Chloramphenicol,Co trimoxazole,Quinolones and Ceftriaxone along with two or more of the following condition

* High grade fever spikes for more than three days
* Refusal to eat or drink
* Drowsy or Unconscious
* Convulsions
* Dehydration due to diarrhea or vomiting
* Abdominal distension with or without tenderness
* Bleeding diathesis like petechial rash, gum bleed, melena
* Jaundice or alanine transaminase more than twice of the normal range
* Thrombocytopenia less than fifty thousand
* Increase Prothrombin time and activated partial thromboplastin time
* Electrolyte imbalance like hyponatremia, hypernatremia, hypokalemia, hyperkalemia, metabolic acidosis
* Hypoglycemia
* Signs of shock like cold and mottled skin, feeble pulses, tachycardia, decreased blood pressure

Exclusion Criteria:

* Not given informed consent
* Children who need ventilator or two inotrope support
* Severe malnutrition/immunocompromised patient

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 126 (Actual)
Dates: Start 2019-06-20 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
clinical clearance | 10 days
  improvement of the signs and symptoms as given in the operational definition

SECONDARY OUTCOMES:
bacterial clearance | 5 days
  negative blood cultures

OTHER OUTCOMES:
relapse of typhoid fever | 15 days after completing treatment
  reappearance of the signs and symptoms of typhoid fever along with positive blood cultures

CONTACTS AND LOCATIONS:
Overall Officials: farhana zafar, mbbs,fcps, Principal Investigator — ziauddin university north campus
Locations (1):
- Ziauddin University, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No